CLINICAL TRIAL: NCT00297804
Title: TAXUS VI - A Randomized, Double-blind Study to Assess Paclitaxel-eluting Stents in Treatment of Longer Lesions
Brief Title: A Randomized, Double-blind Study to Assess Paclitaxel-eluting Stents in Treatment of Longer Lesions
Acronym: TAXUS VI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Thomas Naeschen, Boston Scientific
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2009; TAXUS VI
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Stent Implant; Drug-coated Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Device: TAXUS Express Paclitaxel-Eluting Coronary Stent System
- Arm 2 (Active Comparator)
  Interventions: Device: Control stent

INTERVENTIONS:
Device: TAXUS Express Paclitaxel-Eluting Coronary Stent System — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 1
Device: Control stent — control stent
  Arms: Arm 2

SUMMARY:
The clinical investigation is an international, prospective, multi-center, double-blind, randomized safety and efficacy trial. The purpose of this study is to evaluate the safety and effectiveness of the TAXUS(TM)Stent System with 1µg/mm2 (loaded drug/stent surface area) of paclitaxel incorporated into a moderate rate-release formulation of triblock copolymer carrier system in patients with a higher risk of target lesion revascularisation and restenosis.

DETAILED DESCRIPTION:
The ultimate goal of a paclitaxel eluting stent system is to prevent restenosis by blunting the initial response to stent implant injury and sustaining the arrested response until vascular healing has taken place.

The purpose of the TAXUS VI trial is to study the safety and efficacy of the TAXUS(TM)Stent under controlled trial circumstances and targets patients with a higher risk of target lesion revascularisation and restenosis. The study population will include longer lesions, smaller diameter vessels, multiple lesions in the same vessel, and allows for the use of up to 2 randomized study stents.

The clinical investigation will evaluate the safety and effectiveness of the TAXUS(TM)Stent with 1 µg/mm2 (loaded drug/stent surface area) of paclitaxel incorporated into a moderate rate-release formulation of a triblock copolymer carrier system for treatment of de novo coronary artery lesions.

Patients are stratified by site and presence or absence of medically treated diabetes mellitus and then randomized to receive either the TAXUS(TM)Stent or the uncoated EXPRESS(TM)stent.

The primary objective of the study is to show superior 9-month target vessel revascularization (TVR) rate for TAXUS(TM) Stent compared to uncoated Express(TM)control stent.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria

  1. Patient >or= 18 years old
  2. Eligible for percutaneous coronary intervention
  3. Documented stable angina pectoris or unstable angina pectoris with documented ischemia or documented silent ischemia
  4. Acceptable candidate for CABG
  5. Patient (or legal guardian) understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
  6. Willing to comply with all specified follow-up evaluations
* Angiographic Inclusion Criteria

  1. Target lesion located within a single native coronary vessel
  2. Target lesion randomized to treatment with the study device may be composed of multiple lesions but must be completely coverable by up to 2 study stents (maximum allowable stent length of 48 mm).
  3. Cumulative target lesion length is >or= 18 mm and <or= 40 mm (visual estimate)
  4. RVD of >or= 2.5 mm to <or= 3.75 mm (visual estimate)
  5. Target lesion diameter stenosis >or=50% (visual estimate)
  6. Target lesion is de novo

Exclusion Criteria:

* General Exclusion Criteria:

  1. Known sensitivity to paclitaxel
  2. Any previous or planned treatment with any anti-restenotic drug-coated or drug-eluting coronary stent (Note: previous or planned treatment with heparin or phosphorylcholine coated stents is acceptable, as long as the procedure with the stent meets the protocol defined criteria for staged procedures)
  3. Previous or planned treatment with intravascular brachytherapy in the target vessel
  4. MI within 72 hours prior to the study procedure and/or CK-MB >2x the local laboratory's upper limits of normal (refers to a measured value on the day of the study procedure)
  5. Left ventricular ejection fraction <25%
  6. Cerebrovascular Accident within the past 6 months
  7. Acute or chronic renal dysfunction (creatinine >1.7 mg/dl or >150 µmol/L)
  8. Contraindication to ASA, or to both clopidogrel and ticlopidine
  9. Leukopenia (leukocyte count <3.5 x 109/liter)
  10. Thrombocytopenia (platelet count <100,000/mm3)
  11. Active peptic ulcer or active gastrointestinal bleeding
  12. Known allergy to stainless steel
  13. Any prior true anaphylactic reaction to contrast agents
  14. Known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the study procedure
  15. Patient is currently taking colchicine
  16. Patient is currently, or has been treated with paclitaxel within 12 months of the study procedure
  17. Female of childbearing potential with a positive pregnancy test within 7 days before the study procedure, or lactating, or intends to become pregnant during the study
  18. Life expectancy of less than 24 months due to other medical conditions
  19. Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
  20. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
* Angiographic Exclusion Criteria

  1. Left main coronary artery disease (stenosis >50%), whether protected or unprotected
  2. Target lesion is ostial in location (within 3.0 mm of vessel origin)
  3. Target lesion(s) and/or target vessel proximal to the target lesion(s) is moderately or severely calcified by visual estimation
  4. Target lesion is located within or distal to a >60°bend in the vessel
  5. Target lesion involves a bifurcation with a diseased (>50% stenotic) branch vessel >2.0 mm in diameter
  6. Target lesion is totally occluded Thrombolysis in MI (TIMI flow <or= 1)
  7. Angiographic presence of probable or definite thrombus
  8. Target vessel will be pre-treated with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2002-05; Primary Completion 2003-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Rate of TVR 9 months after index procedure | 9 Months

SECONDARY OUTCOMES:
• Rates of composite Major Adverse Cardiac Events (MACE) and the individual components of MACE, assessed at 1, 3, 6 and 9 months after the study procedure and annually for 5 years (i.e., 1, 2, 3, 4, and 5 years after the study procedure). | 5 years
Stent thrombosis rate. | 5 Years
Target Vessel Failure. | 5 years
Clinical procedural success. | Post procedure
Binary restenosis rate. | 9 months
• Additional angiographic endpoints at 9 month angiographic follow-up | 9 months
IVUS assessment in a subset of approximately 200 patients. At the baseline procedure (post-procedural) and at 9 month follow-up the absolute neointimal volume and the change in neointimal volume from post-procedure to follow-up will be analysed. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, MD, Principal Investigator — HELIOS Clinic Siegburg, Germany
Locations (1):
- HELIOS Clinic, Siegburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wakabayashi K, Mintz GS, Weissman NJ, Stone GW, Ellis SG, Grube E, Ormiston JA, Turco MA, Pakala R, Xue Z, Desale S, Laynez-Carnicero A, Romaguera R, Sardi G, Pichard AD, Waksman R. Impact of drug-eluting stents on distal vessels. Circ Cardiovasc Interv. 2012 Apr;5(2):211-9. doi: 10.1161/CIRCINTERVENTIONS.111.965780. Epub 2012 Apr 10. PMID 22496083